CLINICAL TRIAL: NCT01969760
Title: Pilot-Testing a Family-Based Intervention to Improve Child Outcomes and Increase Family Activity
Acronym: HFDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cassandra Stanton, PhD (Other)
Responsible Party: Sponsor-Investigator, Cassandra Stanton, PhD, Adjunct Assistant Professor of Oncology, Georgetown University
Organization: Georgetown University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-0614
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Smoking; Overweight; Obesity
MeSH Terms: conditions — Smoking; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-list control (No Intervention): Wait-list control. No intervention delivered until post follow-up assessment. Upon completion of the follow-up, the family was offered the full intervention.
- Healthy Families DC Program (Experimental): Healthy Families DC Program
  Interventions: Behavioral: Healthy Families DC Program

INTERVENTIONS:
Behavioral: Healthy Families DC Program — A tailored family-based intervention for health promotion goal setting, substance use prevention, and promotion of physical activity
  Arms: Healthy Families DC Program

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of a family-based program to improve physical activity and tobacco outcomes in a small pilot of middle school students and their families.

DETAILED DESCRIPTION:
Low income ethnic minority youth tend to be at greater risk for obesity, physical inactivity, high risk behaviors such as tobacco and substance use and resulting cardiovascular and chronic disease. In this study we modified a tobacco and substance use risk prevention program to develop a tailored intervention (Healthy Families DC) that also included promotion of physical activity (PA) for DC middle-school students referred by school staff as over-weight and at risk for problem behaviors. The program included an initial family assessment, a family feedback session with family PA goal setting and 6 phone/text based booster sessions. A pilot study with 18 families, comprised of at least one caregiver and target child, was conducted to examine feasibility, acceptability, and trends in preliminary outcomes such as PA via self-report and accelerometry, health risk behaviors (e.g., tobacco use), health goal setting, and changes in family functioning (e.g., youth positive behaviors, parenting).

ELIGIBILITY:
Inclusion Criteria:

* Students aged 12-16 years
* Attending regular education classes at three urban DC public middle schools. -Students must currently reside with at least one parent or guardian who wishes to also participate in this study.
* Students and at least one guardian must be fluent in English

Exclusion Criteria:

* Adolescents, who are outside the study age range
* Patients/parents unable to speak/read English
* Are wards of the state
* Not attending regular education classes at the public middle schools -Furthermore, adolescents and guardians not assenting/consenting to be in the study will be excluded.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Actigraphy-based changes in physical activity from baseline to 8-weeks post-baseline | 8-weeks

SECONDARY OUTCOMES:
Smoking Susceptibility Scale changes from baseline to 8-weeks post-baseline | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra A Stanton, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States